CLINICAL TRIAL: NCT04965662
Title: The Role of Home Packs of HIV Post-Exposure Prophylaxis for Sexual Exposure (PEPSE) to Improve the Speed and Appropriate Uptake of PEPSE in High Risk Individuals
Brief Title: The Role of Home Packs of HIV PEPSE in High Risk Individuals
Acronym: Home PEPSE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: ViiV Healthcare (Industry); Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JF006-3170
Record Dates: First submitted 2021-07-07; First posted 2021-07-16 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — Maraviroc; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Tenofovir; Emtricitabine

STUDY DESIGN:
Intervention Model Description: Individuals at high risk for acquiring HIV will be randomized (1:1) to immediate (ARM A) or deferred (ARM B) Home PEPSE provision (standard of care (SOC)); planned duration of follow-up is 48 weeks for Arm A and 72 weeks for Arm B.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Home PEPSE (Immediate) (Experimental): Patients randomised to the immediate arm (ARM A) will receive a 5 day PEPSE 'Home pack' containing Truvada® (tenofovir disoproxil -as fumarate- 245 mg, emtricitabine 200 mg), ONE tablet OD and Maraviroc 300 mg, TWO tablets OD.
  Interventions: Drug: Maraviroc; Drug: Truvada
- Arm B: Standard of Care (Deferred) (No Intervention): Standard of care antiretroviral therapy for PEPSE as per the British Association for Sexual Health and HIV (BASHH) guidelines.

INTERVENTIONS:
Drug: Maraviroc — Maraviroc 300 mg, TWO tablets once daily.
  Arms: Arm A: Home PEPSE (Immediate)
Drug: Truvada — Truvada one tablet once daily
  Other Names: tenofovir disoproxil -as fumarate- 245 mg, emtricitabine 200 mg
  Arms: Arm A: Home PEPSE (Immediate)

SUMMARY:
The study is looking at a new way to reduce the risk of catching HIV. Post-exposure Prophylaxis for sexual exposure (PEPSE) is where a month of HIV drugs can be given to reduce the chance of getting HIV, after a risk. To improve its use the Investigators want to see whether providing a 5-day course of PEPSE for people to keep at home (HOME PEPSE) will lead to it being taken much quicker than having to get it from sexual health clinics or A&E. The HOME PEPSE packs contain HIV tablets that are used in routine HIV care. However the type of HIV drugs are slightly different to those currently used in PEPSE and the Investigators hope that they will have fewer side effects. HOME PEP consists of Truvada and Maraviroc.

140 gay men who are at high risk of getting HIV will be randomised to one of two groups. Group A will receive HOME PEPSE immediately and group B will receive HOME PEPSE after 48 weeks on the study.

DETAILED DESCRIPTION:
HIV causes significant morbidity and the estimated lifetime cost of one HIV transmission is £0.5-1 million. Despite enormous prevention efforts, transmission rates in the UK remain stable. The population most at risk of acquiring HIV in the UK are men who have sex with men (MSM), who are estimated to number over 500,000 (3.6% of the male population). The estimated prevalence of HIV among MSM aged between 15 and 44 years old is approximately 5%.

In 2013 the highest ever number of new HIV diagnoses (3,000) among MSM was reported and 85% of these were estimated to have been acquired in the UK.

This is supported by a concomitant increase in reported high risk behaviours such as condomless anal sex, from 24.3% to 36.5% of the cohort surveyed in London gyms in 1998 and 2008 respectively. In London, approximately 80% MSM are HIV negative: however high-risk sex continues in the presence of an increasing pool of HIV infected individuals. As such effective HIV prevention interventions are urgently needed to keep such individuals uninfected.

Despite sustained education and public health messages high levels of condomless sex among MSM are reported. HIV prevention tools include condoms, Post-Exposure Prophylaxis following Sexual Exposure (PEPSE), HIV pre-exposure prophylaxis (PrEP), HIV testing to reduce the undiagnosed fraction, antiretroviral treatment (ART) -as-prevention and circumcision. Clinical trials are underway to evaluate the efficacy and cost effectiveness of these approaches.

PEPSE is a key component of HIV prevention. A prospective randomised-controlled trial to determine the efficacy of PEPSE has been precluded due to the high number of participants that would be required for such a study. A case-control study conducted in healthcare workers suggested that the use of zidovudine (AZT) for post exposure prophylaxis after percutaneous exposure to HIV-infected blood was associated with a significant (OR 0.19 (95% CI 0.06-0.52) decrease in the risk of HIV transmission. In addition, mother to child transmission studies where only the neonate received ART have demonstrated a protective effect.

The efficacy of PEPSE is dependent upon the following key factors:

1. Speed of uptake from sexual exposure :

   The time from exposure to initiation of PEPSE is critical for efficacy. Once HIV crosses a mucosal barrier it may take up to 48-72 hours before HIV can be detected within regional lymph nodes and up to five days before HIV can be detected in blood. Initiation of ART has been shown to reduce dissemination and replication of virus in all tissues if initiated early after inoculation in an animal model.

   Animal models mimicking sexual exposure either vaginally or rectally also show protective benefits of the use of ART and demonstrate that time to initiation and duration of PEPSE influence outcome of PEPSE, with delays and shorter courses reducing effectiveness (Tsai J Virol 1998). For example, a phase I/II clinical trial using PMPA (Tenofovir) administered subcutaneously for PEPSE demonstrated that simian immunodeficiency virus (SIV) infection was prevented following an intravenous inoculation in 100% of macaques if administered within 24 hours and continued for 28 days. As either the time to initiation of PEP was increased or the duration of PEPSE was reduced then the number of macaques protected declined.

   Following rectal SIV challenge however, PEPSE offers no protection if taken >24 hours post exposure, with most protection occurring within a 2 hour exposure timeframe. This is of enormous concern for those practicing unprotected receptive anal sex, which is the highest risk sex act for HIV transmission. In the UK, the median time to first PEPSE dose is 24 hours; this unsatisfactory duration has been attributed to the fact that most exposures to HIV occur outside routine clinic hours and a lack of knowledge of where to access PEPSE out-of-hours. Learning from the emergency contraception model women provided with an advance provision of emergency contraception use it to a greater extent and more rapidly after condomless vaginal sex without engaging in increased sexual risk-taking behaviour compared to standard of care.
2. Uptake following sexual exposure. In the Gay Mens survey, 1.7% of gay men reported ever using PEPSE despite 94% reporting at least one sexual partner sex in the preceding year. Approaches to increase PEPSE uptake are therefore required.
3. Adherence

The British Society for Sexual Health and HIV (BASHH) guidelines for PEPSE recommend Truvada and Kaletra for 28 days and the indications for its use are shown in table 1. It is well recognized that ritonavir-boosted protease inhibitors including Kaletra are commonly associated with gastrointestinal side effects and elevations in lipids (Kaletra Spc). Kaletra inhibits cytochrome p450 CYP3A and therefore has many drug-drug interactions. Within the ABT-730 study 37% patients experienced grade 3 or 4 adverse events and laboratory abnormalities in the BD Kaletra arm.

As delayed initiation and non-completion of PEPSE due to side effect are likely to reduce efficacy, it is important to explore regimens that is likely to be better tolerated and ways in which PEPSE could be taken sooner after exposure. Maraviroc (MVC), a CCR5 antagonist has been shown to be an effective antiretroviral agent in the MOTIVATE and MERIT studies. In MERIT the percentage of patients achieving HIV-1 RNA <50 copies/mL was comparable to those receiving efavirenz where they had CCR5-tropic virus at baseline. Maraviroc does not inhibit any of the major P450 enzymes at clinically relevant concentrations (CYP1A2, CYP2B6, CYP2C8, CYP2C9, CYP2C19, CYP2D6 and CYP3A4). Maraviroc appears to have fewer drug-drug interactions than Kaletra and the frequency of grade 3 or 4 adverse events was low (20%) in the MERIT study. Maraviroc acts pre-integration which may have theoretical advantages for PEPSE/PrEP against HIV. Animal data demonstrates that the use of a CCR5 inhibitor reduced the likelihood of macaques acquiring SIV following vaginal exposure. Maraviroc has also been demonstrated to penetrate the male and female genital tract well and achieve high rectal tissue concentrations which may be beneficial for PEP or PrEP. In the event of failure of MVC based PEPSE, it is unlikely treatment options will be affected. Maraviroc is given for HIV treatment twice daily, however safety data supports once daily use and may confer advantages in adherence. Trials evaluating the safety of Maraviroc (MVC) as PEPSE are currently underway in the UK and Spain.

Overall, the cost of PEPSE is minimal in comparison to an HIV transmission and may provide potential cost saving and adherence benefits over daily PrEP. The Investigators propose reducing the time from HIV exposure to first dose of PEPSE in high risk individuals by providing HOME PEPSE (a 5-day pack of PEPSE to be kept at home by the individual in case of need). By removing traditional logistical barriers to PEPSE use, this approach aims to improve the appropriate and immediate access of PEPSE, reduce attendance at A & E, reduce time to first dose (and hence increase efficacy) and further empower individuals to prevent HIV acquisition. If a positive preventative effect is shown then this approach will be evaluated in a large randomised controlled study, rolled out to other NHS providers and is likely to lead to a revision of the UK PEPSE guidelines. Maraviroc lends itself well to episodic, HOME provision PEPSE - it is stable over a long period of time, has fewer drug-drug interactions than protease inhibitors and is well tolerated.

The Investigators hypothesize that advanced provision of PEPSE using Truvada/Maraviroc 600mg OD, so called "HOME" PEPSE to high HIV risk individuals will improve the speed and appropriate uptake of PEPSE and be extremely well tolerated.

140 men who have sex with men and who are at high risk of getting HIV will be randomised to one of two groups. Everyone will be seen at 12 weekly intervals for a sexual behaviour questionnaire and sexual health screen. A more detailed questionnaire will be given at week 0 , week 48 and week 72.

Group A will receive HOME PEPSE immediately and finish the study at week 48. Anyone starting HOME PEPSE will be advised to come to clinic as soon as possible to be assessed for the need for a 28 day PEP course. As starting HOME PEPSE (or standard PEPSE for Arm B) is dependant on participant risk behaviour, HOME PEPSE could not be taken at all during the trial or could be taken multiple times. Therefore how many time certain standard of care/research procedures occur during this trial, such as phlebotomy, is dependant on how many times participants take PEPSE.

Group B will receive HOME PEPSE after 48 weeks on the study and finish the study at week 72. For the first 48 weeks, people in this group will be able to get PEPSE from the normal places i.e. an A&E department or a sexual health clinic. If people do start PEPSE they will be advised to contact the research team so that they can record this and complete a short questionnaire summarizing what happened.

At 48 weeks, everyone will receive a HOME PEPSE pack and have a urine test and blood test to test the kidneys and liver. They will then be followed up for a further 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male gender at birth, age ≥18 years
2. HIV negative by a routinely used assay within 4 weeks prior to or on the day of randomization
3. Willing and able to provide written informed consent
4. And any one of:

   1. condomless anal sex with a male on >1 occasion within the 90 days prior to randomization
   2. bacterial rectal sexually transmitted infection (STI) within the 90 days prior to randomization
   3. use of PEPSE in the 12 months prior to randomization following possible exposure to HIV through unprotected anal intercourse (UAI) with a male

Exclusion Criteria:

1. An acute viral illness that could be due to HIV seroconversion
2. Any contraindications to Truvada or maraviroc according to the current SmPC
3. allergic to soy or peanuts
4. concomitant use of antihypertensive agents
5. history of postural hypotension
6. known hepBsAg positive
7. current participation in a HIV PrEP or PEPSE study
8. Any other active clinically significant condition, or findings during screening medical history or examination, or abnormality on screening laboratory blood tests that would, in the opinion of the investigator, compromise the patient's safety or outcome in the trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 139 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2021-03-16 (Actual)

PRIMARY OUTCOMES:
Number of hours from HIV risk exposure to PEPSE | 48 weeks
  In those accessing PEPSE, the number of hours from HIV sexual risk exposure to initiating PEPSE over 48 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Julie M Fox, MD, Study Director — Chief Investigator-Guy's & St. Thomas' NHS Foundation Trust
Locations (1):
- Guy's & St. Thomas' NHS Foundation Trust, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No